CLINICAL TRIAL: NCT01645020
Title: Comparison Between Two Types of Meshes Used in Pelvic Organs Prolapse Procedures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Postoperative Complications
Keywords: absorbable mesh; Partially absorbed Mesh; Prolift; Prolift + M; mesh related complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Using partially absorbed meshes in pelvic reconstructive surgery will involve fewer postoperative complications especially less pain caused by the mesh mass.

DETAILED DESCRIPTION:
Weakness of pelvic floor support is the cause defects and damage to pelvic organs functioning and urinary control and it has a pretty common occurrence. It was suggested recently that the event is considered a hernia that requires mesh use, which reduces return rates following pelvic floor repair. Mesh use is known to cause complications and unwanted side effects, such as chronic pain, vaginal network exposure and infection. The degree of complications is related directly to the mass of the mesh, and that's why the absorbable meshes were developed.Two months after the surgery with absorbable mesh, the mass left in the patient's body is half of the initial mesh mass and according to our assumption this effect will minimize the extent and intensity of mesh complications compared with conventional ones.

During the study we will examine medical records of women who have had surgery with pelvic floor reconstructive meshes. The cases will be divided according to the mesh type being used.

A polypropylene mesh (single strand and tunneling wide) trade name "Prolift", and similar mesh that contains approximately half of the network mass after being dissolves in two months, a trade name "Prolift +" M.

The number of participants in each group is 120 women. The post-operative follow-up examination will include three points in time. After a month, six months and a year later. In addition to questionnaires in order to quantify the degree of urinary disturbance, pain after surgery and sexual function.

ELIGIBILITY:
Inclusion Criteria:

* Women who had pelvic floor repair surgery wit mesh used to the posterior vaginal wall.

Exclusion Criteria:

* Women with significant pre-operative pain
* Women with collagen diseases
* Women who underwent pelvic floor repair surgery with mesh to the anterior vaginal wall

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: women been operated at Western Galilee Hospital - Nahariya Israel
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2008-08; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: M Neuman, MD, Principal Investigator; Menahem Neuman, Principal Investigator
Locations (1):
- Western Galilee Hospital, Nahariya, Israel

REFERENCES:
- [Background] Khandwala S, Jayachandran C. Transvaginal mesh surgery for pelvic organ prolapse--Prolift+M: a prospective clinical trial. Int Urogynecol J. 2011 Nov;22(11):1405-11. doi: 10.1007/s00192-011-1482-4. Epub 2011 Jul 1. PMID 21720912
- See also: GYNECARE PROLIFT+M™ was developed by Ethicon Women's Health & Urologyoffers. this company offers treatment solutions for a range of female pelvic health disorders. — http://www.ethicon.com/our-story/press-room/prolift_POP_launch